CLINICAL TRIAL: NCT06772051
Title: Short Dentin Etching With a Universal Adhesive: Two-Year Double-Blind Trial Comparing Etching Strategies and Durations
Brief Title: Clinical Evaluation of Short Dentin Etching
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: A04012024 CD
Record Dates: First submitted 2025-01-04; First posted 2025-01-13 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2024-12

CONDITIONS: Hypersensitivity Dentin; Dental Restoration Failure of Marginal Integrity
MeSH Terms: conditions — Dentin Sensitivity

STUDY DESIGN:
Intervention Model Description: Each patient will receive three restorations in posterior teeth randomly on three different quadrants, each tooth will be restored with one of the three tested adhesive strategies. All materials will be used according to manufacturers' instructions
Who Masked: Participant, Investigator
Masking Description: Double (Participant, Investigator)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dentin etching and rinse (15 seconds etching) (Placebo Comparator): The dentin in the pulpal floor in this group will receive phosphoric acid etching for 15 seconds followed by rinsing and drying before universal adhesive application
  Interventions: Procedure: Resin composite restoration bonded using universal adhesive in etch and rinse mode (15 seconds etching)
- Dentin etching and rinse (5 seconds etching) (Active Comparator): The dentin in the pulpal floor in this group will receive phosphoric acid etching for 5 seconds followed by rinsing and drying before universal adhesive application
  Interventions: Procedure: Resin composite restoration bonded using universal adhesive in etch and rinse mode (5 seconds etching)
- Dentin self-etch (Placebo Comparator): The dentin in the pulpal floor in this group will receive universal adhesive application in self-etch mode without prior phosphoric acid etching
  Interventions: Procedure: Resin composite restoration bonded using universal adhesive in self-etch mode

INTERVENTIONS:
Procedure: Resin composite restoration bonded using universal adhesive in etch and rinse mode (15 seconds etching) — Resin composite restoration bonded using universal adhesive in etch and rinse mode (15 seconds etching)
  Arms: Dentin etching and rinse (15 seconds etching)
Procedure: Resin composite restoration bonded using universal adhesive in etch and rinse mode (5 seconds etching) — Resin composite restoration bonded using universal adhesive in etch and rinse mode (5 seconds etching)
  Arms: Dentin etching and rinse (5 seconds etching)
Procedure: Resin composite restoration bonded using universal adhesive in self-etch mode — Resin composite restoration bonded using universal adhesive in self-etch mode
  Arms: Dentin self-etch

SUMMARY:
To evaluate and compare the two-year clinical performance of Class I resin composite restorations utilizing a universal adhesive used in different etch-and-rinse strategies (15-second and 5-second etching) and self-etch strategies for bonding.

DETAILED DESCRIPTION:
The experimental design description adhered to the guidelines provided by the Consolidated Standards of Reporting Trials (CONSORT) statement. The present study is planned as a double-blinded randomized clinical trial, ensuring that both the patients and the examiner are unaware of the treatment allocation. The trial will follow a split mouth design. A total of thirty adult patients, who are seeking dental treatment, will be enrolled in the study. The participants will be recruited from the Operative Department clinic at the Faculty of Dentistry, University of Mansoura. The study will focus on ninety Class I restorations. No active advertisement will be used for participant recruitment, and instead, a convenience sample will be formed. Prior to participating in the study, each patient will be required to provide informed consent by signing a consent form. The study is scheduled to be conducted from December 2024 to December 2026. The form and protocol of the study will be approved by Mansoura University's ethics committee before initiation. To determine the appropriate sample size, previous studies examining the clinical success rate of posterior Class I restorations restored using different adhesive strategies were considered. Based on various parameters, including a significance level of 5%, a test power of 80%, and an equivalence limit of 15%, the sample size was calculated. Considering a potential dropout rate of 20%, a sample size of 30 subjects (Three restorations per patient) was determined to be suitable.

ELIGIBILITY:
Inclusion Criteria:

* Patients with three primary occlusal caries of upper or lower posterior teeth.
* Patients must have a good oral hygiene;
* Patients with tooth gives a positive response to testing with an electric pulp tester
* Patients with normal and full occlusion,
* Patients with opposing teeth should be natural with no restorations.

Exclusion Criteria:

* High caries risk patients with extremely poor oral hygiene

  * Patients involved in orthodontic treatment or periodontal surgery,
  * Patients with periodontally involved teeth (chronic

Ages: 35 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-12-24 (Actual); Primary Completion 2026-12-24 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Postoperative hypersensitivity/pulp status | Two years after restoration
  The postoperative hypersensitivity/pulp status will be assessed based on the updated FDI criteria. This parameter is evaluated by scoring the pain experienced during chewing and/or with cold or warm food items, as reported by the patient. The criteria consist of five scores: scores 1-3 indicate success, score 4 indicates the need for restoration repair, and score 5 indicates the need for restoration replacement.
Marginal adaptation | Two years after restoration
  The marginal adaptation will be evaluated through visual examination using a 250 µm probe and brief air drying. This assessment will be conducted according to the updated FDI criteria. The criteria consist of five scores: scores 1-3 indicate success, score 4 indicates the need for restoration repair, and score 5 indicates the need for restoration replacement.

CONTACTS AND LOCATIONS:
Overall Officials: Hoda S Ismail, Lecturer, Principal Investigator — Faculty of Dentistry, Mansoura University, Egypt
Locations (1):
- Faculty of Dentistry, Mansoura University, Egypt, Al Mansurah, Dakahliya, Egypt